CLINICAL TRIAL: NCT07341997
Title: Environmental Factors Associated With Peripheral Neuropathies in French Guiana
Acronym: YANANER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Admin CIC (Other)
Responsible Party: Sponsor-Investigator, Admin CIC, Nathalie DESCHAMPS, Centre Hospitalier de Cayenne
Organization: Centre Hospitalier de Cayenne (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: YANANER
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Neuropathies; Environmental Risk Factor; Lead Neuropathy; Mercury Neuropathy; Bita
Keywords: Preipheral neuropathies; French guiana; Mercury; Lead; Arboviruses; Environment
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Diagnosis-Related Groups

STUDY DESIGN:
Intervention Model Description: This is a prospective multicenter case-control study being conducted in hospitals in Cayenne and Saint-Laurent du Maroni. At the inclusion visit, blood samples will be taken to assess arbovirus serology, particularly for Zika, Chikungunya and Dengue, as well as to measure levels of heavy metals, including mercury and lead. In addition, urine and hair samples will be taken to analyze these heavy metals. Participants will also fill in a questionnaire about their plant consumption.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control group (Active Comparator): Patients hospitalised or consulting at hospitals in Cayenne and Saint-Laurent du Maroni who do not have peripheral neuropathy.
  Interventions: Other: Case Group

INTERVENTIONS:
Other: Case Group — Patients diagnosed with diabetic peripheral neuropathy or chronic idiopathic axonal polyneuropathy.

SUMMARY:
Peripheral neuropathies (PN) affect 1% of the global population, particularly the elderly. About 20-30% of cases remain unexplained. In French Guiana, we hypothesize that factors like neurotoxic traditional plant remedies, arboviral disease outbreaks, and mercury exposure from illegal gold mining may contribute to PN. The study aims to assess the association between PN and exposure to arboviral infections, heavy metals, and plant consumption in French Guiana.

DETAILED DESCRIPTION:
Peripheral neuropathies (PN) affect 1% of the global population, with higher prevalence in the elderly. They lead to gait disorders and chronic pain, severely impacting quality of life. Despite thorough investigations, 20-30% of cases have no identified cause. In French Guiana, unique factors may contribute to these neuropathies, including the use of potentially neurotoxic traditional plant remedies and outbreaks of arboviral diseases, which can complicate conditions like Guillain-Barré syndrome. Additionally, illegal gold mining exposes residents to mercury, both directly and through environmental contamination. We hypothesize that these local factors might explain the unidentified cases of PN and exacerbate neuropathies in patients with pre-existing nerve vulnerability, such as diabetic neuropathy.

This is a prospective multicenter case-control study being conducted in hospitals in Cayenne and Saint-Laurent du Maroni. At the inclusion visit, blood samples will be taken to assess arbovirus serology, particularly for Zika, Chikungunya and Dengue, as well as to measure levels of heavy metals, including mercury and lead. In addition, urine and hair samples will be taken to analyze these heavy metals. Participants will also fill in a questionnaire about their plant consumption.

They will not be followed as part of the research.

ELIGIBILITY:
Inclusion Criteria:

* For the Case group: patients diagnosed with diabetic peripheral neuropathy or chronic idiopathic axonal polyneuropathy
* For the Control group: patients hospitalized or consulting at the hospitals in Cayenne and Saint-Laurent du Maroni, without peripheral neuropathy.

Exclusion Criteria:

* For the Case and Control groups: patients under the age of 18, those who object to participation and those who are unable to complete the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of exposure rates among cases and controls | At inclusion
  The primary endpoint will be the comparison of rates of exposure to arboviruses, heavy metals and consumption of potentially neurotoxic plants in cases and controls.
  The heavy metals assay and the questionnaire will be carried out at the inclusion visit.

SECONDARY OUTCOMES:
Genetic mutations indentification | At inclusion
  Secondary endpoint will be identification of genetic mutations responsible for peripheral neuropathy
Peripheral Nerve Disability (PND) determination | At inclusion
  Secondary endpoint will be determination of Peripheral Nerve Disability (PND)

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu NACHER, Study Chair — Centre Hospitalier de Cayenne
Locations (2):
- French Guiana (2):
  - Centre Hospitalier de Cayenne, Cayenne
  - Centre Hospitalier de l'Ouest Guyanais, Saint-Laurent-du-Maroni

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nacher M, Ouedraogo E, Succo T, Guarmit B, Djossou F, Stettler L, Alvarez F, Elenga N, Adenis A, Couppié P. L'infection VIH en Guyane: revue historique et tendances actuelles. Bull Epidemiol Hebd. 2020;2-3:43-51. http://beh. santepubliquefrance.fr/beh/2020/2-3/pdf/2020_2-3_2.pdf.
- [Background] Cardoso * T. BA. Le mercure en Guyane française : synthèse des études d'imprégnation et d'impact sanitaires menées de 1994 à 2005. Bulletin Epidémiologique Hebdomadaire - BEH. 2010 Apr;13:118-20.
- [Background] Lernould B. Intoxications à la Bita dans le bassin du Maroni en 2011, série de 4 cas, aspects cliniques et paracliniques, botaniques et de santé publique. Th Doc Méd. Université du Droit et de la Santé - Lille 2, Lille, France. 2013. https://pepite- depot.univ-lille.fr/LIBRE/Th_Medecine/2013/2013LIL2M304. pdf.
- [Background] Graille J, Blaizot R, Darrigade AS, Sainte-Marie D, Nacher M, Schaub R, Couppie P. Leprosy in French Guiana 2007-2014: a re-emerging public health problem. Br J Dermatol. 2020 Jan;182(1):237-239. doi: 10.1111/bjd.18334. Epub 2019 Sep 8. No abstract available. PMID 31286485
- [Background] Sabbah N, Carles G, Demar M, Nacher M. Diabetes in French Guiana, adapting national standards of therapeutic education and care to the amazonian challenge. World J Diabetes. 2021 Feb 15;12(2):98-107. doi: 10.4239/wjd.v12.i2.98. PMID 33594330
- [Background] Maurice L, Barraza F, Blondet I, Ho-A-Chuck M, Tablon J, Brousse P, Demar M, Schreck E. Childhood lead exposure of Amerindian communities in French Guiana: an isotopic approach to tracing sources. Environ Geochem Health. 2021 Nov;43(11):4741-4757. doi: 10.1007/s10653-021-00944-9. Epub 2021 May 11. PMID 33974199
- [Background] Matos LM, Borges AT, Palmeira AB, Lima VM, Maciel EP, Fernandez RNM, Mendes JPL, Romero GAS. Frequency of exposure to arboviruses and characterization of Guillain Barre syndrome in a clinical cohort of patients treated at a tertiary referral center in Brasilia, Federal District. Rev Soc Bras Med Trop. 2022 Apr 8;55:e03062021. doi: 10.1590/0037-8682-0306-2021. eCollection 2022. PMID 35416870
- [Background] Maury-Brachet R, Gentes S, Dassie EP, Feurtet-Mazel A, Vigouroux R, Laperche V, Gonzalez P, Hanquiez V, Mesmer-Dudons N, Durrieu G, Legeay A. Mercury contamination levels in the bioindicator piscivorous fish Hoplias aimara in French Guiana rivers: mapping for risk assessment. Environ Sci Pollut Res Int. 2020 Feb;27(4):3624-3636. doi: 10.1007/s11356-018-3983-x. Epub 2019 Jan 4. PMID 30610584
- [Background] Laperche V, Hellal J, Maury-Brachet R, Joseph B, Laporte P, Breeze D, Blanchard F. Regional distribution of mercury in sediments of the main rivers of French Guiana (Amazonian basin). Springerplus. 2014 Jun 26;3:322. doi: 10.1186/2193-1801-3-322. eCollection 2014. PMID 25045610
- [Background] Schmidt HH, Waddington-Cruz M, Botteman MF, Carter JA, Chopra AS, Hopps M, Stewart M, Fallet S, Amass L. Estimating the global prevalence of transthyretin familial amyloid polyneuropathy. Muscle Nerve. 2018 May;57(5):829-837. doi: 10.1002/mus.26034. Epub 2018 Feb 1. PMID 29211930
- [Background] Pasnoor M, Nascimento OJ, Trivedi J, Wolfe GI, Nations S, Herbelin L, de Freitas MG, Quintanilha G, Khan S, Dimachkie M, Barohn R. North America and South America (NA-SA) neuropathy project. Int J Neurosci. 2013 Aug;123(8):563-7. doi: 10.3109/00207454.2013.782026. Epub 2013 Apr 17. PMID 23461611
- [Background] Hanewinckel R, van Oijen M, Ikram MA, van Doorn PA. The epidemiology and risk factors of chronic polyneuropathy. Eur J Epidemiol. 2016 Jan;31(1):5-20. doi: 10.1007/s10654-015-0094-6. Epub 2015 Dec 23. PMID 26700499